CLINICAL TRIAL: NCT02929927
Title: Acess the Clinical Effect of Antimicrobial Photodynamic Therapy (aPDT) on Root Canal Disinfection
Brief Title: Estimate the Effect of aPDT on Root Canal Disinfection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xiaojing Huang, DDS, PhD, Professor，Vice Dean，School and Hospital of Stomatology Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YTYS83736434
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Root Canal Disinfection
Keywords: Antimicrobial Photodynamic Therapy
MeSH Terms: interventions — Sodium Hypochlorite; Root Canal Preparation; Root Canal Obturation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Experimental): Rubber dam isolation, tooth disinfection，acess to the pulp of the chamber, microbiological sample with two sterile paper points, then mechanical preparation with NITIMTWO to 25#06, and cleaned with 5 ml of 2.5% NaClO between each endodontic file. At the end of the procedure, root canals were ultrasonic irrigated with 2.5% NaClO, 17% EDTA for 1 min followed by irrigation with 0.9% normal saline to remove the smear layer, then take the sample again, drying the canal and fill the canal with a commercial calcium hydroxide-based paste. After 2 weeks, the canals were filled with AH-Plus sealer and Gutta-percha by vertical condensation. The teeth were take crown restoration. Follow up at 3, 6, 12 and 24 months.
  Interventions: Procedure: Rubber dam isolation; Drug: 1% iodine tincture; Drug: 2.5%NaClO; Procedure: root canal preparation; Procedure: root canal obturation
- Experimental group (Experimental): Rubber dam isolation，tooth disinfection，acess to the pulp of the chamber, microbiological sample with two sterile paper points, then mechanical preparation with NITIMTWO to 25#06, and cleaned with 5 ml of 2.5% NaClO between each endodontic file. At the end of the procedure, root canals were ultrasonic irrigated with 2.5% NaClO for 1 min, then 17%EDTA for 1 min followed by irrigation with 0.9% normal saline to remove the smear layer, drying the canal, aPDT, then take the sample again. then dried the canals and filled the canals with AH-Plus sealer and Gutta-percha by vertical condensation. The teeth were take crown restoration. Follow up at 3, 6, 12 and 24 months.
  Interventions: Procedure: Rubber dam isolation; Device: aPDT; Drug: 1% iodine tincture; Drug: 2.5%NaClO; Procedure: root canal preparation; Procedure: root canal obturation

INTERVENTIONS:
Procedure: Rubber dam isolation — tooth was isolated using a rubber dam in order to avoid the outside microbe
Device: aPDT — Inject the photosensitizer (PS)to the parallel orifice of the canal,use the small file to stir the PS for 60 s,then irradiation 120 s.
  Other Names: PADPLUS
  Arms: Experimental group
Drug: 1% iodine tincture — use 1% iodine tincture to disinfect the crown of the teeth.in order to avoid the outside microbe
Drug: 2.5%NaClO — use 2.5% NaClO as irrigants
  Other Names: sodium hypochlorite
Procedure: root canal preparation — mechanical preparation with NITIMTWO to 25#06, and cleaned with 5 ml of 2.5% NaClO between each endodontic file. At the end of the procedure, root canals were ultrasonic irrigated with 2.5% NaClO, 17% EDTA for 1 min followed by irrigation with 0.9% normal saline to remove the smear layer
Procedure: root canal obturation — filled the canals with AH-Plus sealer and Gutta-percha by vertical condensation

SUMMARY:
The aim of this study is to compare the clinical effect of traditional root canal disinfection and aPDT on root canal disinfection. And provide the reference for clinical application and experience.

DETAILED DESCRIPTION:
The study of groups:

Group1: Calcium hydroxide-based antibacterial dressing - two session root canal treatment Group2: aPDT - one session root canal treatment Microbiological measurement. Filled with sterile PBS, the root canals were sampled immediately before and after the disinfection procedures.

ELIGIBILITY:
Inclusion Criteria:

Good general health, without syndromes or chronic systemic diseases; tooth with single root canal; a diagnosis of chronic periapical periodontitis; the lesions of the root tip was less than 6mm; recently (3months)did not take antibiotics.

Exclusion Criteria:

Refused to sign the informed consent document; systemic condition; uncooperative behavior; periodontal-endodontic lesions; allergic to photosensitizer; root apical absorption or destroy; A root canal anatomy of risk factors for the difficulty score ≧ 2

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of bacteria by colony counting | 2 days after the sample taken
  Quantification the total bacteria

SECONDARY OUTCOMES:
tooth pain | 1 week and 3, 6, 12, 24 months after treatment
  patient subjected sensation and doctor remark the symptoms after clinical examination
change of the lesion | 3, 6, 12, 24 months after treatment
  take X ray, measure the lesion and compare to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Huang, PhD, Study Chair — School and Hospital of stomatology,Fujian Medical University
Locations (1):
- School and Hospital of stomatology,Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No